CLINICAL TRIAL: NCT01113593
Title: A Randomized, Multiple-Dose, Crossover Study Characterizing the Pharmacodynamic Profiles of Formoterol Fumarate Inhalation Solution and Formoterol Dry Powder Inhaler in Subjects With Stable Chronic Obstructive Pulmonary Disease
Brief Title: A Study Characterizing Pharmacodynamic Profiles in Subjects With Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dey (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 191-089
Record Dates: First submitted 2010-04-27; First posted 2010-04-30 (Estimated); Last update posted 2013-05-27 (Estimated); Status verified 2013-05

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Formoterol Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Experimental)
  Interventions: Drug: Formoterol Fumarate
- 2 (Experimental)
  Interventions: Drug: Formoterol Fumarate
- 3 (Experimental)
  Interventions: Drug: Formoterol Fumarate
- 4 (Experimental)
  Interventions: Drug: Foradil Aerolizer
- 5 (Experimental)
  Interventions: Drug: Foradil Aerolizer

INTERVENTIONS:
Drug: Formoterol Fumarate — Inhalation solution
  Arms: 1
Drug: Formoterol Fumarate — Inhalation solution
  Arms: 2
Drug: Formoterol Fumarate — Inhalation solution
  Arms: 3
Drug: Foradil Aerolizer — Dry powder inhaler
  Arms: 4
Drug: Foradil Aerolizer — Dry powder inhaler
  Arms: 5

SUMMARY:
The purpose of this study is to characterize the pharmacodynamic profile of Formoterol Fumarate and Foradil Aerolizer

ELIGIBILITY:
Inclusion Criteria:

* Able to understand the requirements of the study and provide informed consent
* A Clinical diagnosis of COPD
* A current or prior history of at least 10-pack years of cigarette smoking
* women of child-bearing potential (WOCBP) must have a negative pregnancy test at the Screening Visit and agree to avoid becoming pregnant for the duration of study

Exclusion Criteria:

* A Clinical Diagnosis of Asthma
* Other significant disease than COPD
* Subjects who radiation or chemotherapy within the previous 12 months
* Subjects who had any lung resection
* QTcB greater than 0.460 seconds
* History of illegal drug abuse or alcohol abuse within the past 5 years

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2010-05; Primary Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Forced expiratory volume at one second (FEV1) measured (in liters) by serial spirometry to compare dosing effect and characterize pharmacodynamic profile of Formoterol Fumarate and Foradil | 12 hours on Day 1 and Day 7 of dosing during each treatment period

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Clearwater, Florida
  - DeLand, Florida
  - Greenville, South Carolina
  - Spartanburg, South Carolina